CLINICAL TRIAL: NCT06817902
Title: A Preliminary Sham-Controlled Theta Burst Stimulation (TBS) Study in Early-Stage Alzheimer's Disease (AD)
Brief Title: TMS Pilot in Early AD II
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A21-251-01
Record Dates: First submitted 2025-02-03; First posted 2025-02-10 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease
Keywords: transmagnetic stimulation; functional MRI guided theta burst stimulation; intermittent theta burst stimulation
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intermittent theta burst stimulation (Experimental): Subjects will receive treatment with intermittent theta burst stimulation (iTBS) with the active coil. There will be a total of 5 treatments over a 2-week period. All subjects will receive iTBS to the 8Av region. TBS treatment will also be provided for two additional sites within the large-scale brain networks (LSBNs) that is found to contain the greatest number of connectivity anomalies. Total participation will be 6-9 weeks.
  Interventions: Device: Intermittent theta burst stimulation active coil
- Sham device (Sham Comparator): Subjects will receive treatment with sham coil. There will be a total of 5 treatments over a 2-week period. Coil will be placed over the same region as the experimental group. Total participation will be 6-9 weeks. An open-label extension will be offered to participants that received the sham (control) treatment without further data collection.
  Interventions: Device: Sham coil

INTERVENTIONS:
Device: Intermittent theta burst stimulation active coil — MagVenture TMS Therapy active coil with theta burst stimulation. Resting motor threshold: 80%; Number of pulses per session: 1200 pulses; Inter-train interval: 8 seconds; Pulse frequency in burst: 50 Hertz
  Other Names: Transmagnetic stimulation; MagVenture
  Arms: Intermittent theta burst stimulation
Device: Sham coil — MagVenture TMS Therapy sham coil
  Other Names: MagVenture
  Arms: Sham device

SUMMARY:
Alzheimer's disease (AD) is a progressive neurodegenerative condition affecting 6.2 million individuals in the United States, resulting in an annual cost of care of $305 billion. AD is functionally characterized by progressive degeneration of large-scale brain networks (LSBNs), including the default mode network (DMN) presumably from the deposition of amyloid plaques and neurofibrillary tangles. Available FDA-approved medications for AD such as donepezil and memantine offer limited benefit and modest impact on quality of life. Transcranial magnetic stimulation (TMS) with intermittent theta burst stimulation (iTBS) offers a non-invasive alternative to pharmacotherapy in persons with AD. We propose a case series study to compare sham with iTBS.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of Mild cognitive impairment (MCI)/mild AD
* Evidence for central nervous system (CNS) amyloidosis (e.g., Amyloid Positron Emission Tomography (PET) or Cerebrospinal fluid (CSF) biomarkers consistent with AD)
* Prior brain imaging performed
* Mini Mental Status Examination (MMSE) >24
* Clinical Dementia Rating (CDR) 0.5-1
* Stable dose of cholinesterase inhibitors and memantine for at least one month
* Subjects are between 40-90 years of age

Exclusion Criteria:

* Non-AD dementia including, but not limited to, Lewy body dementia, frontotemporal dementia, vascular dementia, Jakob-Creutzfeldt disease, etc.
* Inability to tolerate resting state-function magnetic resonance imaging (rs-fMRI)
* Contraindication of rs-fMRI due to implants or metal
* Seizure disorder

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Effect of TBS on cognition between and within subjects using Repeatable Battery for the Assessment of Neuropsychological Status Update (RBANS) | baseline, 7 weeks
  Average change of RBANS total score in TMS arm compared to the average change in RBANS total score in the sham arm. Range [-160 to 160]. Positive comparison of TMS arm to sham arm indicates increased cognitive scores in TMS arm.

CONTACTS AND LOCATIONS:
Overall Officials: Bhavani Kashyap, MBBS, PhD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
No identifiable data will be shared with other researchers.